CLINICAL TRIAL: NCT04782063
Title: Prevention of Obesity in Infants of Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Michael Ross, Distinguished Professor of Obstetrics & Gynecology, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32035-01
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-12

CONDITIONS: Infant Obesity
Keywords: Obesity; Hyperphagia; Breast Milk
MeSH Terms: conditions — Pediatric Obesity; Obesity; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Calibration of infant breast milk and formula intake: We will calibrate (reduce) the pumped breast milk or formula intake of infants of overweight and obese mothers who exceed 75%ile of WHO BMI, in order to prevent infant obesity and subsequent childhood obesity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Standard Infant Feed Group (No Intervention): Infants will receive human milk or formula milk ad libitum.
- Calibrated Infant Feed Group (Other): Infants will have reduced human milk or formula milk intake.
  Interventions: Other: Calibration of infant breast milk and formula milk intake

INTERVENTIONS:
Other: Calibration of infant breast milk and formula milk intake — We will calibrate (reduce) the pumped breast milk or formula intake of infants of overweight and obese mothers who exceed 75%ile of WHO BMI, in order to prevent infant obesity and subsequent childhood obesity.
  Arms: Calibrated Infant Feed Group

SUMMARY:
Maternal and childhood obesity have dramatically increased and continue to present a significant health problem. Studies show that offspring of overweight (body mass index, BMI >25-29.9) and obese (BMI ≥30) women are at increased risk of newborn and age 1-year adiposity, and infant adiposity predicts childhood and adult obesity. The investigators hypothesize that infants of overweight/obese (OW/OB) mothers have both relative hyperphagia and are provided human milk with increased caloric composition, leading to obesity. The investigators propose an intervention study to calibrate milk or formula intake in infants of OW/OB mothers so as to avoid overweight infants at 6 months of age.

DETAILED DESCRIPTION:
This is a clinical intervention study to calibrate infant milk or formula intake and modulate infant weight gain to prevent the development of infant obesity. The investigators will study only OW/OB women, as these patients are at increased risk of infants with excessive weight gain. The study will be conducted using clinical site at Harbor-UCLA Medical Center and at CTSI, The Lundquist Institute.

OW/OB women (pre-pregnant BMI >25-29.9 and ≥30) who are providing exclusive human milk via pumping and bottle (n= 120; 50% male and 50% female) will be recruited postpartum in the hospital or at postpartum visit (typically 3-6 weeks). Study women will be randomly assigned to a Standard Feed (SF) or Calibrated Feed (CF) groups. Mother-infant dyads will be seen at 2-week intervals for assessment of infant milk intake, weight gain, supine length, BMI and skinfold thickness till 6 months of age. Continuation of exclusive human milk will be confirmed with questionnaires.

In the SF group, mothers will provide bottled human milk based upon the volume guidelines: Total daily milk intake recommended will be calculated as infant's weight in ounces divided by 6, with individual feed volume calculated as the total daily volume divided by 6 to 8 (maternal discretion as to number of daily feeds). It is understood that mothers may elect an increased or reduced volume of feed dependent upon infant appetite, behavior, etc. throughout the study, at which time recommended feed volume will be adjusted by the standard formula based upon infant weight.

In the CF group, initial feeding volume will be based upon standard volume guidelines as described above. At the 2 week visits, should infants be within the 75%ile of WHO BMI growth curves, standard weight-based recommended feed volumes will be made. Should the infant be equal or greater than 75%ile of WHO BMI, the recommended human milk feed volume will be reduced by 5% of the weight-based determination, following a consultative assessment by our pediatric/neonatal physician. At subsequent visits, adjustments in human milk volume will continue if the infant exceeds 75%ile of WHO BMI, accommodating the normal increase in human milk intake with advancing weight. In no case, will the daily human milk volume be reduced by more than 10% from the weight-based calculation.

Should the infant be less than 10th percentile of WHO BMI, the maternal-infant dyad will be referred for a pediatric and nutrition consults to assess the cause and treatment for potential nutrient deficiency. At 6 months, the investigators will assess the distribution of infant weight BMI between SF and CF groups.

At the final study visit (6 months), prior to infant feeding, a sample of infant urine will be collected, using the Quick-Wee method with samples collected from voids into plastic bags taped to the genital region. Samples will be analyzed for leptin by ELISA (DLP00, R&D Systems, MN). Urine leptin concentrations correlate significantly with plasma leptin concentration and will provide a non-invasive, semi-quantitative assessment of neonatal hyperleptinemia.

All mothers will quantify and record the daily bottle intake of infants (nearest ml) and will provide a midpumping (8 min) milk sample (10 ml) obtained monthly prior to their visit (morning pumping, frozen) for analysis of protein, carbohydrates and fat (Miris) and total caloric content (bomb calorimetry).

At 6 months, the investigators will assess the distribution of infant weight/BMI between SF and CF groups.

An identical Study (Standard Feed and Calibrated Feed; (n=60 per group; 50% male and 50% female)) will be performed, with the exception that only current formula feed mothers will be enrolled. Daily volume and adjustment of formula feeds will be as described above for human milk. Women will utilize their chosen brand of commercial formula feed, for which total caloric content and composition will be determined.

Data analysis: The proportion of infants whose BMI exceed the 75%ile of WHO BMI at 26 weeks (1st co-primary outcome) will be compared between the two group (SF vs CF) using a pooled z-test or Fisher's exact test. Growth curves for SF and CF over 26 weeks will be estimated and the area under the curve (AUC) compared with the 75%ile curve of WHO BMI. AUCs (secondary outcome) will be computed using the trapezoidal method or integrations of the estimated closed form of the mathematical function. The difference between these AUCs represents the magnitude of how long and much BMI exceed the 75%ile of WHO BMI over the 6 month period. These AUC between the two groups will be compared using a two sample t-test. As exploratory analyses, if potential covariates are found, multivariate analyses (linear and generalized linear regression models) will be used to adjust confounding effects. Sub-group analyses will be also carried out, such as by gender. The investigators will also investigate if early changes in growth curves or maternal human milk composition are associated with infant weight changes, so as to determine the potential for invention prior to exceeding the 75%ile of WHO BMI.

ELIGIBILITY:
Inclusion Criteria:

* Breast Milk Calibration Study: Study women (pre-pregnant BMI 25-29.9 and ≥30) who are providing exclusive human milk via pumping and bottle (50%/50% male/female) will be recruited at the 3-6 week postpartum visit.
* Formula Milk Calibration Study: Study women (pre-pregnant BMI 25-29.9 and ≥30) who are providing formula via bottle (50%/50% male/female) will be recruited at the 3-6 week postpartum visit.

Exclusion Criteria:

* Breast Milk Calibration Study: breast implants, prior breast surgery, flat/ inverted nipples, tongue-tie or low birth weight infants.
* Formula Milk Calibration Study: low birth weight infants.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Infant normalized weight at 6 months of age | 6 months
  We will quantify effects of calibrated human milk or formula intake on the normalized weight of infants at 6 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Ross, MD, Principal Investigator — Lundquist Institute
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at national and international meetings spanning obstetrics, pediatrics and public health. The findings of the study will be published according to NIH guideline for publication and accepted manuscripts will be deposited to Pub Med Central to ensure public access.
  For the community, we will disseminate research data through educational program, workshops and conferences organized by The Lundquist Institute. It is important to note that we plan to translate our research findings into Spanish.
Supporting Information: CSR
Time Frame: Data available at completion of protocol estimated Nov 2023
Access Criteria: Established research organization

REFERENCES:
- [Background] Brunner S, Schmid D, Zang K, Much D, Knoeferl B, Kratzsch J, Amann-Gassner U, Bader BL, Hauner H. Breast milk leptin and adiponectin in relation to infant body composition up to 2 years. Pediatr Obes. 2015 Feb;10(1):67-73. doi: 10.1111/j.2047-6310.2014.222.x. Epub 2014 Apr 14. PMID 24729519
- [Result] Satpathy HK, Fleming A, Frey D, Barsoom M, Satpathy C, Khandalavala J. Maternal obesity and pregnancy. Postgrad Med. 2008 Sep 15;120(3):E01-9. doi: 10.3810/pgm.2008.09.1920. PMID 18824817
- [Result] Kaul P, Bowker SL, Savu A, Yeung RO, Donovan LE, Ryan EA. Association between maternal diabetes, being large for gestational age and breast-feeding on being overweight or obese in childhood. Diabetologia. 2019 Feb;62(2):249-258. doi: 10.1007/s00125-018-4758-0. Epub 2018 Nov 13. PMID 30421138
- [Result] Davenport MH, Cabrero MR. Maternal nutritional history predicts obesity in adult offspring independent of postnatal diet. J Physiol. 2009 Jul 15;587(Pt 14):3423-4. doi: 10.1113/jphysiol.2009.174896. No abstract available. PMID 19602635
- [Result] Guo SS, Wu W, Chumlea WC, Roche AF. Predicting overweight and obesity in adulthood from body mass index values in childhood and adolescence. Am J Clin Nutr. 2002 Sep;76(3):653-8. doi: 10.1093/ajcn/76.3.653. PMID 12198014
- [Result] Catalano PM. Obesity and pregnancy--the propagation of a viscous cycle? J Clin Endocrinol Metab. 2003 Aug;88(8):3505-6. doi: 10.1210/jc.2003-031046. No abstract available. PMID 12915626
- [Result] Prentice P, Ong KK, Schoemaker MH, van Tol EA, Vervoort J, Hughes IA, Acerini CL, Dunger DB. Breast milk nutrient content and infancy growth. Acta Paediatr. 2016 Jun;105(6):641-7. doi: 10.1111/apa.13362. Epub 2016 Apr 6. PMID 26865238
- [Result] Isganaitis E, Venditti S, Matthews TJ, Lerin C, Demerath EW, Fields DA. Maternal obesity and the human milk metabolome: associations with infant body composition and postnatal weight gain. Am J Clin Nutr. 2019 Jul 1;110(1):111-120. doi: 10.1093/ajcn/nqy334. PMID 30968129
- [Result] Young BE, Levek C, Reynolds RM, Rudolph MC, MacLean P, Hernandez TL, Friedman JE, Krebs NF. Bioactive components in human milk are differentially associated with rates of lean and fat mass deposition in infants of mothers with normal vs. elevated BMI. Pediatr Obes. 2018 Oct;13(10):598-606. doi: 10.1111/ijpo.12394. Epub 2018 Aug 9. PMID 30092608